CLINICAL TRIAL: NCT06586099
Title: Prospective, Open-label, Single Arm Trial to Evaluate Efficacy and Safety of Tislelizumab with Azacitidine in the Treatment of Refractory/relapsed Acute Myeloid Leukemia
Brief Title: Tislelizumab with Azacitidine in the Treatment of R/R AML
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: withdrawn
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020007
Record Dates: First submitted 2020-07-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Refractory AML; Relapsed Adult AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: prospective, open label, single arm clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): azacytidine 75mg/m2/d, IH,day1-7, every 28 days for three cycles tislelizumab 200mg,day 8,every three weeks, for 4 doses
  Interventions: Drug: Aza, tislelizumab

INTERVENTIONS:
Drug: Aza, tislelizumab — combination chemotherapy for the refractory/relapsed AML

SUMMARY:
Acute myeloid leukemia(AML) is a clonal hematological malignancy. 50%-90% adult AML patients can achieve complete remission(CR) after standard induction chemotherapy,but 10%-25% patients cannot achieve CR, which is called 'primary refractory disease'.Most of patients who achieved CR will relapse during the next 3 years, and the prognosis is poor.So refractory and relapse diseases are still the hotspot of clinical research.Immunologic escape is one of the mechanisms for tumor cells to survive from chemotherapy. Studies have shown that PD1 and PDL1 levels are upregulated in AML patients, the same phenomenon was observed after the treatment of demethylating agents such as azacytidine. Combination of PD1 blockades with azacytidine may improve the efficacy of the treatment.

DETAILED DESCRIPTION:
In this phase 1/2 study, 20 patients will be enrolled and treated with azacytidine and tislelizumab regimen. The primary endpoint is composite complete remission rate.Toxicities of treatment need to be observed. And relationship between PDL1 expression on AML cells and efficacy will be studied. Treatments include azacytidine 75mg/m2/d, subcutaneous injection,day1-7, every 28 days for three cycles tislelizumab 200mg,day 8,every three weeks, for 4 doses.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of AML according to FAB or WHO criteria
* refractory or morphological relapsed AML
* age over 18 years old
* ECOG PS 0-2
* written informed consent

Exclusion Criteria:

* acute promyelocyte leukemia
* solitary extramedullary relapsed disease
* other hematological diseases
* antecedent stem cell transplantation
* AML with BCR_ABL positive
* acute panmyelosis with myelofibrosis or sarcoma
* with other active organ malignancy(needing treatment)
* active heart diseases
* unfit for enrollment after investigator's evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
composite complete remission rate | up to 2 years
  including complete remission plus complete remission with incomplete blood cell count recovery

SECONDARY OUTCOMES:
overall survival | up to 4 years
  The interval from the date of enrollment to the date of death or the date of last follow-up, whichever occurred first.
disease free survival | up to 4 years
  From CR1 to relapse, death from any cause or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- HBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No